CLINICAL TRIAL: NCT06357065
Title: Effectiveness of the Active Transport Educational Program Based on the Ecological Model on Improving the Physical and Mental Health of Secondary Students: Study Protocol for a Randomized Controlled Trial (Mov-Es Project)
Brief Title: Active Transport Educational Program Based on the Ecological Model on Improving the Physical and Mental Health: MOV-ES Project
Acronym: MOV-ES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Eugenio Merellano Navarro, Research Associate, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UCatolicaMaule; 11240343 (Other Grant/Funding Number: ANID Chile)
Record Dates: First submitted 2024-03-27; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity in Children
Keywords: physical activity; active transport; schoolchildren
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Study design, setting: This is a cluster randomized field trial aimed to evaluate the previously tested MOV-ES intervention.
  Population: First year of high school students in a city in south-central Chile. Three secondary schools in the urban area of Talca (1 public, 1 private subsidized, and 1 private non-subsidized) with at least three classes per school year will be randomly selected. This methodological option was adopted because, in Chile, school administration is associated with the socioeconomic level of families.
Who Masked: Investigator
Masking Description: Randomization and blinding procedures: We invited 6 first-year high school classes to participate and, using a computer-generated procedure, will be randomized to the IG and to CG. The participants will be informed of the result of randomization after they agreed to participate in the study. The nature of the intervention makes its blinding infeasible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOV-ES group (Experimental): The design of the intervention requires incorporating content that involves intrapersonal (benefits of active transportation and safety on the way to school), interpersonal (family safety), organizational, community, physical-environmental, and political (safety, infrastructure, quality) factors. It will consist of weekly sessions of 60 to 90 minutes each for 16 weeks. The complete program has a duration of 4 months, during school hours in the subject of Physical Education, and on the premises of each establishment. The contents to be worked on will be organized in a Didactic Unit and will include the presentation of graphic and audiovisual material and practical contents. Each session will be designed based on the results of PHASE 1 of the study, following the recommendations of active transport interventions in schoolchildren , and the material available from the PACO Project.
  Interventions: Other: Active transport educational program based on the ecological model
- Control group (No Intervention): The CG students will participate in the initial and final measurement, but will not receive any intervention, attending their traditional Physical Education classes.

INTERVENTIONS:
Other: Active transport educational program based on the ecological model — The intervention is structured according to the following units: Unit I: benefits of physical activity on health and healthy habits in schoolchildren; Unit II: Active Transportation: Experiences from other countries; Unit III: Analysis of the environmental characteristics of the school environment of each establishment; and Unit VI: Road safety for pedestrians and cyclists. This last topic will be broken down considering analysis and prevention of accidents with automobiles, pedestrian regulations, signaling, and cyclist safety. The sessions of the last month of intervention (November) will include practical walking activities in the school environment (outside the school). Depending on the possibilities of each school, cycling sessions will be included.
  Arms: MOV-ES group

SUMMARY:
The epidemic of physical inactivity affects the entire world and is responsible for more than 5 million deaths per year. The call of the United Nations, through the 2030 Agenda and the Sustainable Development Goals, encourages the creation of favorable environments for physical activity based on the ecological model of physical activity. Given this context, active transportation can be an accessible, economical, and sustainable method to increase daily physical activity. The rate of school children who use active transport has decreased, being replaced by motorized transport, causing congestion and high levels of pollution in cities. In the Chilean context, there are studies of active transportation in the Chilean population; however, they are scarce in the school population and none of them is an intervention study, demonstrating the incipient development of this area in the country. The benefits of promoting active transportation not only favor the lifestyles of school children but also include additional co-benefits such as the improvement of mental health and better academic performance, in addition to the reduction of exhaust and greenhouse gas emissions.

Objectives. This proposal consists of three phases with the following objectives: Phase I: i) to synthesize the evidence about interventions aimed at estimating the effect on health of active transport in the secondary students; and ii), using qualitative techniques, to explore, from the basis of grounded theory, barriers and facilitators perceived by professors, students and parents about the development and implementation of the MOV-ES intervention. Phase II. Pilot and feasibility trial: a) to test the effect of MOV-ES intervention on improving body composition (body fat percentage and muscle mass), physical fitness (aerobic capacity and muscular strength), executive function and mental fitness (mood disorders, cognitive functioning) in the secondary students; and b), to examine the acceptability by professors, parents and students of the intervention by using ad hoc questionnaires. Phase III: to test the effectiveness of the MOV-ES intervention on physical activity, physical fitness, cognition and mental health through a cluster randomized controlled trial.

Expected results: This project will give rise to the following master's and doctoral theses, with their corresponding articles of high scientific impact: 1) Barriers and facilitators of teachers, parents and students for active transport from a qualitative approach; 2) Association between the built environment, urban features, and active transportation in high school students, 3) Effectiveness of an active transportation educational intervention on physical fitness and body composition, 4) Effectiveness of an active transportation educational intervention on the cognition of schoolchildren. It is expected that the results of the MOV-ES Project will transcend the physical health of schoolchildren and will have an impact on the school community, especially by decongesting the school environment. Through these results, the Ministry of Education, regional DAEM, municipalities, and educational establishments will be able to propose public policies that favor the practice of physical activity and the acquisition of healthy habits at school age. All of the above is based on quality indicators proposed by the Education Quality Agency.

ELIGIBILITY:
Inclusion Criteria:

* Students in their third year of high school enrolled in schools in the province of Talca

Exclusion Criteria:

* Students who have some motor problem to carry out autonomous transportation.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Body composition change (fat mass) by bioimpedance at 16 weeks | 4 months
  The body composition (bioimpedance), the percentage of fat mass will be obtained using eight electrode tetrapolar bioimpedance (InBody 570®, Body Composition Analyzers, South Korea).
Change from Body Composition (fat-free mass) by bioimpedance at 16 weeks | 4 months
  The body composition (bioimpedance), the percentage of fat-free mass will be obtained using eight electrode tetrapolar bioimpedance (InBody 570®, Body Composition Analyzers, South Korea). Score Test d'Dimensional Chang Card Sort Test Score Test d'List Sorting Working Memory Test
Changes in Executive Function (inhibition) at 16 weeks | 4 months
  Inhibitory control and attention will be measured using the Flaker Attention and Inhibitory Control Test (NIH Toolbox). The participant is asked to focus on a particular stimulus while inhibiting attention to the stimuli flanking it. By applying the test, a score of inhibitory control and attention is obtained.
Changes in Executive Function (cognitive flexibility) at 16 weeks | 4 months
  Cognitive flexibility and attention will be measured using the Dimensional Change Card Sort Test (NIH Toolbox). The participant is asked to match a series of picture pairs to a target picture. A score of cognitive flexibility and attention is obtained by applying the test.
Changes in executive function (working memory) at 16 weeks | 4 months
  Working memory will be measured using list sorting working memory test. Test available at NIH Toolbox. The participant is asked to recall and sequence different stimuli that are presented visually and via audio. A working memory score is obtained by applying the test

SECONDARY OUTCOMES:
Change from Anthropometric measurements at 16 weeks | 4 months
  The following anthropometric measurements will be obtained: i) body weight in kg with a digital scale (Seca 769, Germany; Accuracy of 0.1 kg); ii) bipedal height in cm with a stadiometer (Seca 220, Germany; Accuracy of 0.1 cm). Weight and height will be combined to report BMI in kg/m^2.
Changes in objective physical activity at 16 week | 4 months
  Measurement of objective physical activity will be by Actigraph Accelerometer - Model wGT3X-BT. They include a microelectromechanical system (MEMS) based accelerometer, ambient light and a touch sensor as data collection endpoints. The study subjects will wear the device for 6 full days. The analysis of the data extracted from the accelerometers will allow to identify and classify the amount (minutes) of physical activity performed according to its intensity (low, moderate and high).
Change from Physical Fitness (Aptitud cardiorrespiratoria (VO2 máx) at 16 weeks | 4 months
  VO2 max will be measured using the 20m shuttle run test, , which allows for a highly reliable and easy-to-use evaluation. . This is a maximal test involving a continuous run between two lines separated by 20 m at the same time as the beeps are recorded. The athlete's score is the level and number of laps (20 m) achieved before he/she could not keep up with the recording. The level score can be converted to an equivalent VO 2max score.
Change from Physical Fitness (lower body strength) at 16 weeks | 4 months
  Lower body strength will be measured using the feet together long jump test, which allows for a highly reliable and easy-to-use evaluation. Test to measure or assess the explosive force (power) of the tensor muscles of the legs. The number of centimeters advanced, from the jump line to the edge closest to the jump line, of the foot that was farthest behind after the fall is recorded. The distance in centimeters becomes a power category.
Change from Physical-Functional Fitness (strenght on the upper body) at 16 weeks | 4 months
  This will be evaluated with the hydraulic dynamometer (Camry, model EH101, China), which allows evaluation of great reliability and easy application. The arm curl test to assess the strength on the upper body, using a 3lb (women) and 5lb (men) dumbbell, counting the number of repetitions made in 30s.
Change from mental health (depression) at 16 weeks | 4 months
  This will be evaluated with the Depression, Anxiety, and Stress Scale (DASS-21). Is an instrument designed to assess the negative emotional states of depres-sion, anxiety, and stress. The depression subscale formed by questions 3, 5, 10, 13, 16, 17, and 21. The total scores cate-gorize each subscale into three levels: mild, mo-derate, and severe. Finally, participants will be classified as no risk (<6) or risk (>6).
Change from mental health (Anxiety) at 16 weeks | 4 months
  This will be evaluated with the Depression, Anxiety, and Stress Scale (DASS-21). Is an instrument designed to assess the negative emotional states of depres-sion, anxiety, and stress. Questions 2, 4, 7, 9, 15, 19, and 20 formed the anxiety subscale. The total scores cate-gorize each subscale into three levels: mild, mo-derate, and severe. Finally, participants will be classified as no risk (<6) or risk (>6).
Change from mental health (Stress) at 16 weeks | 4 months
  This will be evaluated with the Depression, Anxiety, and Stress Scale (DASS-21). Is an instrument designed to assess the negative emotional states of depres-sion, anxiety, and stress. The stress subscale was formed by questions 1, 6, 8, 11, 12, 14, and 18. The total scores cate-gorize each subscale into three levels: mild, mo-derate, and severe. Finally, participants will be classified as no risk (<6) or risk (>6).
Changes in overall academic performance once the intervention is completed | 5 months
  To evaluate this variable, the grades of all subjects from the first academic semester will be considered and compared with that of the second semester (intervention). The rating scale in Chile is from 1 to 7, with 7 being the maximum rating.
Changes in health-related quality of life at 16 weeks | 4 months
  This will be obtained using the Kidscreen-52, which measures the attributes of ten dimensions of health: Physical well-being, Psychological well-being, Moods and emotions, Self-perception, Autonomy, Relationships with parents and home life, Financial resources, Peers and social support, School Environment, Bullying. Each dimension is made up of a series of questions that together give a scale ranging from 0 (the worst health state for that dimension) to 100 (the best health state).
Changes in the Perception of urban environmental characteristics at 16 weeks | 4 months
  To measure the Perception of environmental urban features, the Neighborhood environment walkability scale questionnaire was used. (NEWS). It measures the following eight walkability constructs using 66 questions: residential density, land use mix, access to land use mix, street connectivity, walking and biking infrastructure, aesthetics, safety/traffic hazards and security against crime. Additionally, the questionnaire has questions about individual satisfaction with the neighborhood. Higher scores mean greater perception of the urban environment to promote active transportation.
Changes in physical activity barriers at 16 weeks | 4 months
  The Short scale of perception of barriers for physical activity in adolescents will be used. Twelve-item self-report instrument that asks adolescents to declare to what extent they perceive the different items included in the scale as barriers to not practicing organized sports activities. Each item was assessed with a five-point Likert-type response scale in which 1 means totally disagree and 5 means totally agree.
Changes in adherence to physical activity at 16 weeks | 4 months
  The Physical Activity Questionnaire for Adolescents (PAQ-A) will be completed. Self-report scale, described by its creators as designed for use with scalar students, contains eight items intended to capture adolescents' recall of their physical activity during the previous 7 days. The first and last of the eight items of the PAQ-A each contain a number of sub-items from which a mean is initially calculated, and these two means are added to the responses of the other six items to obtain a total a from which the mean is calculated to produce a composite score ranging from 1 to 5, with higher scores indicating greater PA.Puntuación del examen
Changes in the form of Transportation to and from School (Active Transportation) at 16 weeks. | 4 months
  The questions of the questionnaire will be used based on the PACO Project. The question will be directly asked about the way in which you travel to and from school in the last week. The response options are: Motorized transportation, by bicycle and walking.

OTHER OUTCOMES:
Sociodemographic evaluations of parents | 2 weeks
  Age (years), academic level (primary, secondary, bachelor, master, PhD), civil status (married, separated, widow, single, others).
Parents' perception of urban environmental characteristics | 2 weeks
  To measure the Perception of urban environmental characteristics, the neighborhood environmental walkability scale questionnaire was used. (NEWS parent version). Measures the following eight walkability constructs using 66 questions: residential density, land use mix, access to land use mix, street connectivity, walking and biking infrastructure, aesthetics, safety/traffic hazards, and security against crime. Additionally, the questionnaire has questions about individual satisfaction with the neighborhood. Higher scores mean greater awareness of the urban environment to promote active transportation.
Parents' perception of physical fitness | 2 weeks
  Parents' Self-Perceived Physical Condition Level The International Fitness Scale (IFIS) will be used. Instrument composed of five questions on a Likert scale that ask about the general fitness perceived by adults (general physical condition, respiratory physical condition, strength, speed/agility and flexibility in comparison with physical fitness with people of the same age (very poor, bad, average, good and very good).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohl HW 3rd, Craig CL, Lambert EV, Inoue S, Alkandari JR, Leetongin G, Kahlmeier S; Lancet Physical Activity Series Working Group. The pandemic of physical inactivity: global action for public health. Lancet. 2012 Jul 21;380(9838):294-305. doi: 10.1016/S0140-6736(12)60898-8. PMID 22818941
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Aubert S, Barnes JD, Abdeta C, Abi Nader P, Adeniyi AF, Aguilar-Farias N, Andrade Tenesaca DS, Bhawra J, Brazo-Sayavera J, Cardon G, Chang CK, Delisle Nystrom C, Demetriou Y, Draper CE, Edwards L, Emeljanovas A, Gaba A, Galaviz KI, Gonzalez SA, Herrera-Cuenca M, Huang WY, Ibrahim IAE, Jurimae J, Kamppi K, Katapally TR, Katewongsa P, Katzmarzyk PT, Khan A, Korcz A, Kim YS, Lambert E, Lee EY, Lof M, Loney T, Lopez-Taylor J, Liu Y, Makaza D, Manyanga T, Mileva B, Morrison SA, Mota J, Nyawornota VK, Ocansey R, Reilly JJ, Roman-Vinas B, Silva DAS, Saonuam P, Scriven J, Seghers J, Schranz N, Skovgaard T, Smith M, Standage M, Starc G, Stratton G, Subedi N, Takken T, Tammelin T, Tanaka C, Thivel D, Tladi D, Tyler R, Uddin R, Williams A, Wong SHS, Wu CL, Zembura P, Tremblay MS. Global Matrix 3.0 Physical Activity Report Card Grades for Children and Youth: Results and Analysis From 49 Countries. J Phys Act Health. 2018 Nov 1;15(S2):S251-S273. doi: 10.1123/jpah.2018-0472. PMID 30475137
- [Background] Guthold R, Stevens GA, Riley LM, Bull FC. Worldwide trends in insufficient physical activity from 2001 to 2016: a pooled analysis of 358 population-based surveys with 1.9 million participants. Lancet Glob Health. 2018 Oct;6(10):e1077-e1086. doi: 10.1016/S2214-109X(18)30357-7. Epub 2018 Sep 4. PMID 30193830
- [Background] Aguilar-Farias N, Miranda-Marquez S, Martino-Fuentealba P, Sadarangani KP, Chandia-Poblete D, Mella-Garcia C, Carcamo-Oyarzun J, Cristi-Montero C, Rodriguez-Rodriguez F, Delgado-Floody P, Von Oetinger A, Balboa-Castillo T, Pena S, Cuadrado C, Bedregal P, Celis-Morales C, Garcia-Hermoso A, Cortinez-O'Ryan A. 2018 Chilean Physical Activity Report Card for Children and Adolescents: Full Report and International Comparisons. J Phys Act Health. 2020 Jul 15;17(8):807-815. doi: 10.1123/jpah.2020-0120. Print 2020 Aug 1. PMID 32668409
- [Background] Celis-Morales C, Salas C, Martinez MA, Leiva AM, Garrido-Mendez A, Diaz-Martinez X. [The economic burden of physical inactivity in Chile]. Rev Med Chil. 2017 Aug;145(8):1091-1092. doi: 10.4067/s0034-98872017000801091. No abstract available. Spanish. PMID 29189871
- [Background] Aznar S, Naylor PJ, Silva P, Perez M, Angulo T, Laguna M, Lara MT, Lopez-Chicharro J. Patterns of physical activity in Spanish children: a descriptive pilot study. Child Care Health Dev. 2011 May;37(3):322-8. doi: 10.1111/j.1365-2214.2010.01175.x. Epub 2010 Nov 18. PMID 21083695
- [Background] Stanley RM, Maher C, Dollman J. Modelling the contribution of walking between home and school to daily physical activity in primary age children. BMC Public Health. 2015 May 1;15:445. doi: 10.1186/s12889-015-1765-7. PMID 25928079
- [Background] Costa J, Adamakis M, O'Brien W, Martins J. A Scoping Review of Children and Adolescents' Active Travel in Ireland. Int J Environ Res Public Health. 2020 Mar 18;17(6):2016. doi: 10.3390/ijerph17062016. PMID 32197539
- [Background] Aarts MJ, Mathijssen JJ, van Oers JA, Schuit AJ. Associations between environmental characteristics and active commuting to school among children: a cross-sectional study. Int J Behav Med. 2013 Dec;20(4):538-55. doi: 10.1007/s12529-012-9271-0. PMID 23076641
- [Background] Kek CC, Garcia Bengoechea E, Spence JC, Mandic S. The relationship between transport-to-school habits and physical activity in a sample of New Zealand adolescents. J Sport Health Sci. 2019 Sep;8(5):463-470. doi: 10.1016/j.jshs.2019.02.006. Epub 2019 Feb 28. PMID 31534821
- [Background] Martin A, Boyle J, Corlett F, Kelly P, Reilly JJ. Contribution of Walking to School to Individual and Population Moderate-Vigorous Intensity Physical Activity: Systematic Review and Meta-Analysis. Pediatr Exerc Sci. 2016 Aug;28(3):353-63. doi: 10.1123/pes.2015-0207. Epub 2016 Feb 17. PMID 26882871
- [Background] Salvo D, Garcia L, Reis RS, Stankov I, Goel R, Schipperijn J, Hallal PC, Ding D, Pratt M. Physical Activity Promotion and the United Nations Sustainable Development Goals: Building Synergies to Maximize Impact. J Phys Act Health. 2021 Jul 13;18(10):1163-1180. doi: 10.1123/jpah.2021-0413. PMID 34257157
- [Background] Sarmiento OL, Lemoine P, Gonzalez SA, Broyles ST, Denstel KD, Larouche R, Onywera V, Barreira TV, Chaput JP, Fogelholm M, Hu G, Kuriyan R, Kurpad A, Lambert EV, Maher C, Maia J, Matsudo V, Olds T, Standage M, Tremblay MS, Tudor-Locke C, Zhao P, Church TS, Katzmarzyk PT. Relationships between active school transport and adiposity indicators in school-age children from low-, middle- and high-income countries. Int J Obes Suppl. 2015 Dec;5(Suppl 2):S107-14. doi: 10.1038/ijosup.2015.27. Epub 2015 Dec 8. PMID 27152178
- [Background] Martin-Moraleda E, Mandic S, Queralt A, Romero-Blanco C, Aznar S. Associations among Active Commuting to School and Prevalence of Obesity in Adolescents: A Systematic Review. Int J Environ Res Public Health. 2022 Aug 31;19(17):10852. doi: 10.3390/ijerph191710852. PMID 36078573
- [Background] Andersen LB, Wedderkopp N, Kristensen P, Moller NC, Froberg K, Cooper AR. Cycling to school and cardiovascular risk factors: a longitudinal study. J Phys Act Health. 2011 Nov;8(8):1025-33. doi: 10.1123/jpah.8.8.1025. PMID 22039135
- [Background] Larouche R, Saunders TJ, Faulkner G, Colley R, Tremblay M. Associations between active school transport and physical activity, body composition, and cardiovascular fitness: a systematic review of 68 studies. J Phys Act Health. 2014 Jan;11(1):206-27. doi: 10.1123/jpah.2011-0345. Epub 2012 Dec 17. PMID 23250273
- [Background] Fromel K, Groffik D, Mitas J, Dygryn J, Valach P, Safar M. Active Travel of Czech and Polish Adolescents in Relation to Their Well-Being: Support for Physical Activity and Health. Int J Environ Res Public Health. 2020 Mar 18;17(6):2001. doi: 10.3390/ijerph17062001. PMID 32197391
- [Background] Carver A, Salmon J, Campbell K, Baur L, Garnett S, Crawford D. How do perceptions of local neighborhood relate to adolescents' walking and cycling? Am J Health Promot. 2005 Nov-Dec;20(2):139-47. doi: 10.4278/0890-1171-20.2.139. PMID 16295706
- [Background] Rodriguez-Rodriguez F, Cristi-Montero C, Celis-Morales C, Escobar-Gomez D, Chillon P. Impact of Distance on Mode of Active Commuting in Chilean Children and Adolescents. Int J Environ Res Public Health. 2017 Nov 2;14(11):1334. doi: 10.3390/ijerph14111334. PMID 29099044
- [Background] Gonzalez SA, Sarmiento OL, Lemoine PD, Larouche R, Meisel JD, Tremblay MS, Naranjo M, Broyles ST, Fogelholm M, Holguin GA, Lambert EV, Katzmarzyk PT. Active School Transport among Children from Canada, Colombia, Finland, South Africa, and the United States: A Tale of Two Journeys. Int J Environ Res Public Health. 2020 May 28;17(11):3847. doi: 10.3390/ijerph17113847. PMID 32481728
- [Background] Salvo D, Reis RS, Sarmiento OL, Pratt M. Overcoming the challenges of conducting physical activity and built environment research in Latin America: IPEN Latin America. Prev Med. 2014 Dec;69 Suppl 1:S86-92. doi: 10.1016/j.ypmed.2014.10.014. Epub 2014 Oct 16. PMID 25456800
- [Background] McDonald NC. Active transportation to school: trends among U.S. schoolchildren, 1969-2001. Am J Prev Med. 2007 Jun;32(6):509-16. doi: 10.1016/j.amepre.2007.02.022. PMID 17533067
- [Background] Dalton MA, Longacre MR, Drake KM, Gibson L, Adachi-Mejia AM, Swain K, Xie H, Owens PM. Built environment predictors of active travel to school among rural adolescents. Am J Prev Med. 2011 Mar;40(3):312-9. doi: 10.1016/j.amepre.2010.11.008. PMID 21335262
- [Background] Garcia-Hermoso A, Hormazabal-Aguayo I, Fernandez-Vergara O, Gonzalez-Calderon N, Russell-Guzman J, Vicencio-Rojas F, Chacana-Canas C, Ramirez-Velez R. A before-school physical activity intervention to improve cognitive parameters in children: The Active-Start study. Scand J Med Sci Sports. 2020 Jan;30(1):108-116. doi: 10.1111/sms.13537. Epub 2019 Sep 2. PMID 31410887
- [Background] Chaddock-Heyman L, Erickson KI, Voss MW, Knecht AM, Pontifex MB, Castelli DM, Hillman CH, Kramer AF. The effects of physical activity on functional MRI activation associated with cognitive control in children: a randomized controlled intervention. Front Hum Neurosci. 2013 Mar 12;7:72. doi: 10.3389/fnhum.2013.00072. eCollection 2013. PMID 23487583
- [Background] Sallis JF, Cervero RB, Ascher W, Henderson KA, Kraft MK, Kerr J. An ecological approach to creating active living communities. Annu Rev Public Health. 2006;27:297-322. doi: 10.1146/annurev.publhealth.27.021405.102100. PMID 16533119
- [Background] Sarmiento OL, Rubio MA, King AC, Serrano N, Hino AAF, Hunter RF, Aguilar-Farias N, Parra DC, Salvo D, Jauregui A, Lee RE, Kohl B. Built environment in programs to promote physical activity among Latino children and youth living in the United States and in Latin America. Obes Rev. 2021 Jun;22 Suppl 3(Suppl 3):e13236. doi: 10.1111/obr.13236. Epub 2021 Apr 6. PMID 33825294
- [Background] Ding D, Sallis JF, Conway TL, Saelens BE, Frank LD, Cain KL, Slymen DJ. Interactive effects of built environment and psychosocial attributes on physical activity: a test of ecological models. Ann Behav Med. 2012 Dec;44(3):365-74. doi: 10.1007/s12160-012-9394-1. PMID 22899301
- [Background] Cerin E, Conway TL, Cain KL, Kerr J, De Bourdeaudhuij I, Owen N, Reis RS, Sarmiento OL, Hinckson EA, Salvo D, Christiansen LB, Macfarlane DJ, Davey R, Mitas J, Aguinaga-Ontoso I, Sallis JF. Sharing good NEWS across the world: developing comparable scores across 12 countries for the Neighborhood Environment Walkability Scale (NEWS). BMC Public Health. 2013 Apr 8;13:309. doi: 10.1186/1471-2458-13-309. PMID 23566032
- [Background] Adams MA, Frank LD, Schipperijn J, Smith G, Chapman J, Christiansen LB, Coffee N, Salvo D, du Toit L, Dygryn J, Hino AA, Lai PC, Mavoa S, Pinzon JD, Van de Weghe N, Cerin E, Davey R, Macfarlane D, Owen N, Sallis JF. International variation in neighborhood walkability, transit, and recreation environments using geographic information systems: the IPEN adult study. Int J Health Geogr. 2014 Oct 25;13:43. doi: 10.1186/1476-072X-13-43. PMID 25343966
- [Background] Santos MP, Page AS, Cooper AR, Ribeiro JC, Mota J. Perceptions of the built environment in relation to physical activity in Portuguese adolescents. Health Place. 2009 Jun;15(2):548-552. doi: 10.1016/j.healthplace.2008.08.006. Epub 2008 Sep 20. PMID 19004663
- [Background] Sallis JF, Spoon C, Cavill N, Engelberg JK, Gebel K, Parker M, Thornton CM, Lou D, Wilson AL, Cutter CL, Ding D. Co-benefits of designing communities for active living: an exploration of literature. Int J Behav Nutr Phys Act. 2015 Feb 28;12:30. doi: 10.1186/s12966-015-0188-2. PMID 25886356
- [Background] Larouche R, Mammen G, Rowe DA, Faulkner G. Effectiveness of active school transport interventions: a systematic review and update. BMC Public Health. 2018 Feb 1;18(1):206. doi: 10.1186/s12889-017-5005-1. PMID 29390988
- [Background] Bustos N, Olivares S, Leyton B, Cano M, Albala C. Impact of a school-based intervention on nutritional education and physical activity in primary public schools in Chile (KIND) programme study protocol: cluster randomised controlled trial. BMC Public Health. 2016 Dec 3;16(1):1217. doi: 10.1186/s12889-016-3878-z. PMID 27912741
- [Background] Cruz TH, Davis SM, Myers OB, O'Donald ER, Sanders SG, Sheche JN. Effects of an Obesity Prevention Intervention on Physical Activity Among Preschool Children: The CHILE Study. Health Promot Pract. 2016 Sep;17(5):693-701. doi: 10.1177/1524839916629974. Epub 2016 Apr 18. PMID 27091603
- [Background] Ramanathan S, O'Brien C, Faulkner G, Stone M. Happiness in motion: emotions, well-being, and active school travel. J Sch Health. 2014 Aug;84(8):516-23. doi: 10.1111/josh.12172. PMID 25040120
- [Background] Martinez-Gomez D, Ruiz JR, Gomez-Martinez S, Chillon P, Rey-Lopez JP, Diaz LE, Castillo R, Veiga OL, Marcos A; AVENA Study Group. Active commuting to school and cognitive performance in adolescents: the AVENA study. Arch Pediatr Adolesc Med. 2011 Apr;165(4):300-5. doi: 10.1001/archpediatrics.2010.244. Epub 2010 Dec 6. PMID 21135316
- [Background] Hagel BE, Macpherson A, Howard A, Fuselli P, Cloutier MS, Winters M, Richmond SA, Rothman L, Belton K, Buliung R, Emery CA, Faulkner G, Kennedy J, Ma T, Macarthur C, McCormack GR, Morrow G, Nettel-Aguirre A, Owens L, Pike I, Russell K, Torres J, Voaklander D, Embree T, Hubka T. The built environment and active transportation safety in children and youth: a study protocol. BMC Public Health. 2019 Jun 11;19(1):728. doi: 10.1186/s12889-019-7024-6. PMID 31185992
- [Background] de Nazelle A, Nieuwenhuijsen MJ, Anto JM, Brauer M, Briggs D, Braun-Fahrlander C, Cavill N, Cooper AR, Desqueyroux H, Fruin S, Hoek G, Panis LI, Janssen N, Jerrett M, Joffe M, Andersen ZJ, van Kempen E, Kingham S, Kubesch N, Leyden KM, Marshall JD, Matamala J, Mellios G, Mendez M, Nassif H, Ogilvie D, Peiro R, Perez K, Rabl A, Ragettli M, Rodriguez D, Rojas D, Ruiz P, Sallis JF, Terwoert J, Toussaint JF, Tuomisto J, Zuurbier M, Lebret E. Improving health through policies that promote active travel: a review of evidence to support integrated health impact assessment. Environ Int. 2011 May;37(4):766-77. doi: 10.1016/j.envint.2011.02.003. PMID 21419493
- [Background] Garrido-Mendez A, Diaz X, Martinez MA, Leiva AM, Alvarez C, Ramirez Campillo R, Cristi-Montero C, Rodriguez F, Salas-Bravo C, Duran E, Labrana AM, Aguilar-Farias N, Celis-Morales C. [Association of active commuting with obesity: findings from the Chilean National Health Survey 2009-2010]. Rev Med Chil. 2017 Jul;145(7):837-844. doi: 10.4067/s0034-98872017000700837. Spanish. PMID 29182191
- [Background] Herreros-Irarrazabal D, Guzman-Habinger J, Mahecha Matsudo S, Kovalskys I, Gomez G, Rigotti A, Cortes LY, Yepez Garcia MC, Pareja RG, Herrera-Cuenca M, Farias-Valenzuela C, Marques A, Leme ACB, Fisberg M, Drenowatz C, Ferrari G. Association between Active Transportation and Public Transport with an Objectively Measured Meeting of Moderate-to-Vigorous Physical Activity and Daily Steps Guidelines in Adults by Sex from Eight Latin American Countries. Int J Environ Res Public Health. 2021 Nov 3;18(21):11553. doi: 10.3390/ijerph182111553. PMID 34770064
- [Background] Garcia-Hermoso A, Saavedra JM, Olloquequi J, Ramirez-Velez R. Associations between the duration of active commuting to school and academic achievement in rural Chilean adolescents. Environ Health Prev Med. 2017 Apr 4;22(1):31. doi: 10.1186/s12199-017-0628-5. PMID 29165126
- [Background] Mandic S, Williams J, Moore A, Hopkins D, Flaherty C, Wilson G, Garcia Bengoechea E, Spence JC. Built Environment and Active Transport to School (BEATS) Study: protocol for a cross-sectional study. BMJ Open. 2016 May 24;6(5):e011196. doi: 10.1136/bmjopen-2016-011196. PMID 27221127
- [Background] Dimaggio C, Li G. Effectiveness of a safe routes to school program in preventing school-aged pedestrian injury. Pediatrics. 2013 Feb;131(2):290-6. doi: 10.1542/peds.2012-2182. Epub 2013 Jan 14. PMID 23319533
- [Background] Villa-Gonzalez E, Ruiz JR, Chillon P. Associations between Active Commuting to School and Health-Related Physical Fitness in Spanish School-Aged Children: A Cross-Sectional Study. Int J Environ Res Public Health. 2015 Aug 26;12(9):10362-73. doi: 10.3390/ijerph120910362. PMID 26322487
- [Background] Villa-Gonzalez E, Ruiz JR, Ward DS, Chillon P. Effectiveness of an active commuting school-based intervention at 6-month follow-up. Eur J Public Health. 2016 Apr;26(2):272-6. doi: 10.1093/eurpub/ckv208. Epub 2015 Nov 16. PMID 26578663
- [Background] Buliung R, Faulkner G, Beesley T, Kennedy J. School travel planning: mobilizing school and community resources to encourage active school transportation. J Sch Health. 2011 Nov;81(11):704-12. doi: 10.1111/j.1746-1561.2011.00647.x. PMID 21972991
- [Background] Ducheyne F, De Bourdeaudhuij I, Lenoir M, Cardon G. Effects of a cycle training course on children's cycling skills and levels of cycling to school. Accid Anal Prev. 2014 Jun;67:49-60. doi: 10.1016/j.aap.2014.01.023. Epub 2014 Feb 4. PMID 24607594
- [Background] Coombes E, Jones A. Gamification of active travel to school: A pilot evaluation of the Beat the Street physical activity intervention. Health Place. 2016 May;39:62-9. doi: 10.1016/j.healthplace.2016.03.001. Epub 2016 Mar 11. PMID 26974232
- [Background] Cabanas-Sanchez V, Tejero-Gonzalez CM, Veiga OL. [Construction and validation of a short scale of perception of barriers for the physical activity in adolescents]. Rev Esp Salud Publica. 2012 Jul-Aug;86(4):435-43. doi: 10.4321/S1135-57272012000400010. Spanish. PMID 23076088
- [Background] Martinez-Gomez D, Gomez-Martinez S, Warnberg J, Welk GJ, Marcos A, Veiga OL. Convergent validity of a questionnaire for assessing physical activity in Spanish adolescents with overweight. Med Clin (Barc). 2011 Jan 15;136(1):13-5. doi: 10.1016/j.medcli.2010.05.013. Epub 2010 Aug 10. PMID 20701933
- [Background] Ortega FB, Ruiz JR, Espana-Romero V, Vicente-Rodriguez G, Martinez-Gomez D, Manios Y, Beghin L, Molnar D, Widhalm K, Moreno LA, Sjostrom M, Castillo MJ; HELENA study group. The International Fitness Scale (IFIS): usefulness of self-reported fitness in youth. Int J Epidemiol. 2011 Jun;40(3):701-11. doi: 10.1093/ije/dyr039. Epub 2011 Mar 24. PMID 21441238
- See also: Global school-based student health survey — https://www.who.int/teams/noncommunicable-diseases/surveillance/systems-tools/global-school-based-student-health-survey